CLINICAL TRIAL: NCT03478488
Title: Gemcitabine and Oxaliplatin With or Without KN035 for Biliary Tract Cancer: a Randomised, Open-label, Parallel-group, Multicenter Phase III Study
Brief Title: Programmed Death Ligand (PD-L1) Combined With Chemotherapy for Patients With BTC
Acronym: KN035-BTC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: 3D Medicines (Sichuan) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: 3D Medicines (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KN035-CN-005
Record Dates: First submitted 2018-03-21; First posted 2018-03-27 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Biliary Tract Neoplasms
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — envafolimab; Gemcitabine; Oxaliplatin; gemcitabine-oxaliplatin regimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KN035 (Experimental): KN035 plus Gemcitabine & oxaliplatin KN035 2.5 mg/Kg, administered as subcutaneous injection, weekly of each 21-day cycle.
  Gemcitabine 1000 mg/m^2, IV infusion on Day 1 and Day 8, and oxaliplatin 85 mg/m^2, IV infusion on Day 1 of each 21-day cycle for no more than 6 cycles.
  Interventions: Drug: KN035 plus Gemcitabine & oxaliplatin
- Gemcitabine & oxaliplatin (Active Comparator): Gemcitabine 1000 mg/m^2, IV infusion on Day 1 and Day 8, and oxaliplatin 85 mg/m^2, IV infusion on Day 1 of each 21-day cycle for no more than 6 cycles.
  Interventions: Drug: Gemcitabine & oxaliplatin

INTERVENTIONS:
Drug: KN035 plus Gemcitabine & oxaliplatin — KN035 a programmed death ligand immune check inhibitor Per Investigator decision
  Other Names: Experimental
  Arms: KN035
Drug: Gemcitabine & oxaliplatin — The standard of care for the patients with unresectable/metastatic biliary tract cancer
  Other Names: Active Comparator
  Arms: Gemcitabine & oxaliplatin

SUMMARY:
This is a randomized, open-label, parallel-group multi-center study of Phase 3 study to assess the efficacy and safety of KN035 compared to standard of care (SOC) Gemcitabine-based chemotherapies in the treatment of participants with previously untreated locally advanced or metastatic biliary tract cancer.

The primary hypothesis of this study is that participants will have a longer overall Survival (OS) when treated with combined therapy than SOC.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years and older;
* Histological or cytological diagnosis of unresectable or metastatic gallbladder cancer or cholangiocarcinoma;
* Previously untreated with systemic therapy; Subjects who developed recurrent disease >6 months after a sort of adjuvant, neoadjuvant chemotherapy could also be eligible.
* Liver function Child-Pugh A or B;
* Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status;
* Life expectancy of at least 12 weeks;
* At least one measurable lesion per RECIST 1.1;
* Adequate organ function

Exclusion Criteria:

* Specific anti-tumor treatment prior to 4 weeks;
* more than 50% liver metastasis ;
* Patient with other serious diseases or clinical conditions, including but not limited to uncontrolled active infection etc;
* History of severe hypersensitivity reaction to any monoclonal antibody or chemistry;
* Women who are pregnant or in the period of lactation;
* Patients with an active, known or suspected autoimmune disease. Patients are permitted to enrol if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2018-04-16 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Observed by 12 weeks after progressive disease or end of treatment
  was defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Observed by 6 weeks
  was defined as the time from randomization to documented disease progression per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) or death due to any cause, whichever occurred first and was based on blinded independent Review Committee (BIRC) review.
Objective response rate (ORR) | Observed by 6 weeks
  was defined as the percentage of participants in the analysis population who experienced a Complete Response or a Partial Response and was assessed using RECIST 1.1 based on BIRC evaluation.
Disease control rate (DCR) | Observed by 6 weeks
  was defined as the percentage of participants in the analysis population who experienced a Complete Response or a Partial Response or stable disease and was assessed using RECIST 1.1 based on BIRC evaluation
Duration of Response (DOR) | Observed by 6 weeks
  was defined as the time from the first met for complete response/partial response (whichever was first recorded) until the first date that recurrent or progressive disease was objectively documented (taking as reference for progressive disease the smallest measurements recorded on study)
Time to progression (TTP) | Observed by 6 weeks
  was defined as the time from randomization to the first date that progressive disease was objectively documented

CONTACTS AND LOCATIONS:
Overall Officials: Shukui Qin, Principal Investigator — The Chinese people's liberation army (PLA) 81 hospital
Locations (1):
- The Chinese people's liberation army (PLA) 81hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided